CLINICAL TRIAL: NCT06524388
Title: The Effects of COgNitive Training in Community-dwelling Older Adults at High Risk for demENTia and With Diabetes (CONTENT-Diabetes): a Randomized, Placebo-controlled Trial
Brief Title: Adaptive Cognitive Training on Cognitive Function in Elderly Diabetes Patients in the Community
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fanfan Zheng (Other)
Responsible Party: Sponsor-Investigator, Fanfan Zheng, Principal Investigator, Peking Union Medical College
Organization: Peking Union Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CFH 2024-2G-4253
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-02

CONDITIONS: Cognition; Diabetes Mellitus, Type 2; Aging
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adaptive cognitive training (Experimental): The intervention lasted for 12 weeks. Participants will revieve 30 minutes of training per day, at least five days per week. In each task, once a high accuracy (e.g. >80%) is achieved, the task is automatically upgraded to the next difficulty level.
  Interventions: Device: adaptive cognitive training
- placebo cognitive training (Placebo Comparator): The intervention lasted for 12 weeks. Participants will revieve 30 minutes of training per day, at least five days per week. The tasks will be set to a fixed level of difficulty.
  Interventions: Device: placebo cognitive training

INTERVENTIONS:
Device: adaptive cognitive training — The intervention was computerized, multi-domain, adaptive cognitive training. Training areas include processing speed, attention, perception, long-term memory, working memory, computation, executive control, reasoning, and problem-solving. Embedded in the Adaptive Cognitive training application is an adaptive algorithm that will help provide each participant with a cognitive training task at the right level of difficulty based on their profile and real-time performance.
  Arms: adaptive cognitive training
Device: placebo cognitive training — Participants received cognitive training tasks of fixed difficulty.
  Arms: placebo cognitive training

SUMMARY:
Objective A growing body of evidence supports diabetes as a risk factor for cognitive decline. Diabetes is significantly associated with accelerated cognitive decline, poorer cognitive function, and mild cognitive impairment and dementia. Cognitive training is an effective intervention to improve cognitive function. However, the current cognitive training does not fully consider the different areas and degrees of cognitive function impairment of older adults. This study aims to evaluate the effect of adaptive cognitive training on cognitive function of older adults with hypertension in the community.

Participants Age 60 years or older, diagnosis of diabetes, fasting blood glucose≥6.1mmol/L and cognitive function assessment showed no dementia.

Design The study was designed as a double-blind randomized controlled trial. 120 diabetes participants without dementia aged 60 years or older in Shijingshan, Beijing and Haidian, Beijing were included. Participants will be randomized to adaptive cognitive training (intervention group) and placebo cognitive training (control group) at a ratio of 1:1. Both training will be delivered by using PADs with the same appearance. The interventions will last for 6 months and follow up to 12 months, and both groups will be followed up on the same time schedules for all outcome measurements. The primary outcome is changes in MoCA scores from baseline to post-intervention, 6 months. The current trial has been reviewed by the Ethics Committee of Plastic Surgery Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College (approval number: 2024-162).

ELIGIBILITY:
Inclusion Criteria:

* with a clear diagnosis of diabetes (according to ICD-10 or DSM-criteria), fasting blood glucose≥6.1mmol/L, maintaining the original diabetes treatment strategy
* age ≥60 years old
* literate and able to use smart phone or tablet computer skillfully, with CAIDE dementia risk score >9, but without a diagnosis of dementia (ICD-10 or DSM-dementia diagnostic criteria)
* have lived in the target community for at least 6 months and continue to live in the original community for the next 12 months

Exclusion Criteria:

* Stroke or brain surgery in the previous 12 months
* Alcohol or drug abuse in the past 12 months
* Families, important people of participants in the study have concerns
* Live in the same household as a participant who has been randomly assigned
* Severe aphasia, physical disability, or any other factor that may prevent completion of neuropsychological testing
* Use of medications that may affect cognition, including sedatives, anxiolytics, hypnotics, nootropics, and cholinergic drugs; Refusing or not receiving cognitive training
* currently participating in another clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | baseline; "post-intervention, 12weeks"
  MoCA has been widely used in the cognitive function assessment of middle-aged and elderly people in China, including executive function, memory, orientation, computation, conceptual thinking, visual perception, language, and attention. The MoCA scale scores ranged from 0 to 30, and the lower the score, the worse the cognitive function.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | baseline; 6 week-intervention; "post-intervention, 12 weeks"; 24 weeks follow-up
  MoCA has been widely used in the cognitive function assessment of middle-aged and elderly people in China, including executive function, memory, orientation, computation, conceptual thinking, visual perception, language, and attention. The MoCA scale scores ranged from 0 to 30, and the lower the score, the worse the cognitive function.
the Trail Making Test (TMT) | baseline; 6 week-intervention; "post-intervention, 12 weeks"; 24 weeks follow-up
  The TMT assesses cognitive processing speed and executive function. The TMT consists of two parts, A and B, and is one of the most widely used neuropsychological assessment tools. The TMT-A requires the subject to connect disorderly arranged numbers from 1 to 25 in order. Investigator used a modified version that included numbers in both square and circle figures and required participants to alternate the two figures when connecting the numbers in order. The score index was the time spent on TMT-A and TMT-B and the amount of interference (time spent on TMT-B - time spent on TMT-A).
the Digit Symbol Substitution Test (DSST) | baseline; 6 week-intervention; "post-intervention, 12 weeks"; 24 weeks follow-up
  DSST has 1-9 numbers and corresponding symbols. Subjects were required to correctly fill in the symbols under the numbers according to the corresponding relationship between numbers and symbols in the 90s content. One point was calculated for every one completed within 90 seconds, and the higher the score, the better the cognitive function.
the WHO-UCLA Auditory Verbal Learning Test(AVLT) | baseline; 6 week-intervention; "post-intervention, 12 weeks"; 24 weeks follow-up
  AVLT consisted of 15 words, which were read aloud at a rate of one word in 2 seconds while the subject listened. After reading aloud, the subjects were asked to recall the words as much as possible for 90 seconds, and the recall did not have to be in the order of reading aloud. During the recall process, the examiner recorded the correct words and their number, inserted and repeated words. The above reading and immediate recall were repeated 5 times. The total score of AVLT recall from 1 to 5 passes was the total score of immediate recall. Delayed recall and cued recall were also performed, and distractor exclusion recall was performed.
the Boston Naming Test (BNT) | baseline; 6 week-intervention; "post-intervention, 12 weeks"; 24 weeks follow-up
  There were 30 pictures in the BNT, and subjects were required to name the pictures, each of which was scored on a scale of 0-2. Two points were given for complete correctness, one point for semantic errors, and zero points for other situations. The sum of the scores of all objects gives a total score, with a maximum score of 60.
Geriatric Depression Scale (GDS) | baseline; 6 week-intervention; "post-intervention, 12 weeks"
  GDS describes the participant's depressive symptoms in the past week on a scale of 0 to 15, with higher scores indicating more severe depressive symptoms.
Generalized Anxiety Disorder-7 (GAD-7) | baseline; 6 week-intervention; "post-intervention, 12 weeks"
  GAD-7 assesses the anxiety of the participants in the past two weeks, with a total of 7 items. The total score ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Pittsburgh sleep quality index (PSQI) | baseline; 6 week-intervention; "post-intervention, 12 weeks"
  PSQI assesses the subjective sleep quality of participants in the past month. The total score ranges from 0 to 21, with higher scores indicating worse sleep quality.
fasting blood glucose | baseline; "post-intervention, 12 weeks"
  Fasting blood glucose will be obtained by blood samples,which will be collected by nurses from community hospitals in a fasted state (at least 8 hours without food or water).

CONTACTS AND LOCATIONS:
Locations (1):
- Xihuangcun Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Trial outcome data and essential baseline characteristics data are available upon request. Researchers interested in accessing the trial dataset should contact the corresponding author with details of their proposed research use. Data access will be provided subject to review and approval of the research protocol and execution of a data use agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Pan Y, Ji M, Liang J, Ma J, Zhang W, Liu Y, Dai Y, Gao D, Zhang Y, Xie W, Zheng F. Effects of COgNitive Training in Community-dwelling Older Adults at High Risk for demENTia (CONTENT): study protocol of two double-blind, randomised, placebo-controlled trials. BMJ Open. 2026 Feb 9;16(2):e095515. doi: 10.1136/bmjopen-2024-095515. PMID 41663164